CLINICAL TRIAL: NCT06863025
Title: Effects of Neurofeedback Training on Attentional Deficits in Patients With Acquired Brain Injury
Acronym: NeMoRe
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Hospitales Nisa (Other)
Collaborators: Horizon 2020 - European Commission (Other)
Responsible Party: Principal Investigator, Enrique Noe, Dr, Hospitales Nisa
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: NeMoRe
Record Dates: First submitted 2024-10-11; First posted 2025-03-07 (Actual); Last update posted 2025-03-07 (Actual); Status verified 2024-09

CONDITIONS: Brain Injuries; Attention Disorder
Keywords: neurofeedback; brain injury; attentional deficits; neuromodulation; neurorehabilitation
MeSH Terms: conditions — Brain Injuries; Cognition Disorders

STUDY DESIGN:
Intervention Model Description: two groups: 1)experimental will receive treatment (NF), 2) control will receive standard cognitive therapy rehabilitation. groups will be matched for numbers of treatment received
Who Masked: Outcomes Assessor
Masking Description: data will be coded and anonymised before performing the analyses on the outcome measures
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Neurofeedback (Experimental): This group will receive 12 sessions of neurofeedback (20 minutes each session) targeting beta and theta. The neurofeedback protocol will aim at increasing frequencies between 16-25 and decreasing 4-7 Hz
  Interventions: Behavioral: Neurofeedback training
- Control (Active Comparator): This group will receive 12 sessions of standard practice cognitive therapy (20 minutes each session) targeting attentional deficits.
  Interventions: Behavioral: Standard cognitive therapy

INTERVENTIONS:
Behavioral: Neurofeedback training — Neurofeedback (NF) or electroencephalographic feedback (EEG) training refers to a type of computerized cognitive training that changes EEG patterns through operant conditioning. NF is a computerized rehabilitation technique but also a non-invasive neuromodulation approach, as it alters brain activity by delivering a stimulus. It is well-established for the treatment of conditions such as anxiety and ADHD. During NF rehabilitative training, the subject is provided with real-time EEG feedback, usually with a visual or auditory stimulus, with the aim of normalizing brain oscillations. Rehabilitation through NF training generally targets EEG frequencies that are affected and underlie the observed behavioral deficit (e.g., attentional dysfunctions).
  Arms: Neurofeedback
Behavioral: Standard cognitive therapy — This is the control intervention and it involves standard practice cognitive therapy in neurorehabilitation. Neuropsychologists and other clinicians test and train the patients' cognitive specific aspect (in this case, attention) with some validated tools and/or games
  Arms: Control

SUMMARY:
The goal of this study is to investigate new neuromodulation therapies for attention deficits following acquired brain injury. Brain damage can affect various domains, including motor and cognitive functions. However, cognitive deficits have many consequences on the functionality and independence of patients, and attention is an essential requirement for most of daily activities. After brain damage, cognitive rehabilitation is generally the first treatment option for attention deficits. Some studies have shown that cognitive rehabilitation is sometimes not very effective.

For this reason, new therapies such as neuromodulation techniques are being investigated. Neurofeedback is a non-invasive neuromodulation therapy involving a type of computer-based training and learning, and some studies have shown that it is a promising tool to treat cognitive deficits in patients with brain injuries.

In the present study, the investigators will evaluate the effects of neurofeedback as a therapy for attentional deficits after brain injury. Participants undergoing neurofeedback and cognitive therapy will be compared to participants only receiving cognitive therapy.

ELIGIBILITY:
Inclusion Criteria:

* ≥18 years old
* ABI resulting from TBI, stroke, hypoxia and other etiologies
* attentional deficits that are among the objectives of neurorehabilitation as established by the clinical team (scores falling in the 90% percentiles on the Conner's Continuous Performance - CCPT, on the Digit and Spatial Span Tasks and Color Trail test)
* good cognitive condition (ie., scores of ≥23 in the Mini Mental State Examination
* MMSE or ≥75 in the Galveston Orientation & Amnesia Test - GOAT)

Exclusion Criteria:

* previous report of psychiatric and/or neurologic disorders
* contraindication to computerized activities
* blindness or severe visual impairments

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2024-10-01 (Actual); Primary Completion 2025-06-30 (Estimated); Study Completion 2025-10-01 (Estimated)

PRIMARY OUTCOMES:
Behavioral effectiveness of NF on attention measures - CCPT | The CCPT will be assessed during the pre-treatment assessment (within three weeks before the start of the treatment) and the post-treatment assessment (within 3 weeks of the end of the treatment)
  The Conners Continuous Performance Test (CCPT ) is a computer administered test designed to assess problems with attention. It presents 360 stimuli trials (i.e., individual letters) on the screen, with 1, 2, or 4 seconds intervals between the presentation. The 360 trials are divided into 18 blocks of 20 trials each and participants instructed to press the spacebar or the appropriate key on the mouse for any letter that appears, except the letter "X." The CCPT takes 14 minutes to administer. Through the various measures of the CCPT we can measure different aspects of attentional deficits such as processing speed, sustained and selective attention, inhibition, vigilance, inattention.
Behavioral effectiveness of NF on attention measures - Color Trail Test | The Color Trail Test will be assessed during the pre-treatment assessment (within three weeks before the start of the treatment) and the post-treatment assessment (within 3 weeks of the end of the treatment)
  The Color Trail Test evaluates processing speed, selective attention, sequencing, mental flexibility, visual search, and motor function. It has been used for detecting cognitive impairment in early stages and a wide variety of neurological processes and disorders. In Part A of the test, the subject is presented with a sheet with numbers from 1 to 25 placed inside circles and distributed randomly across an A4-sized sheet. The task involves connecting the numbers consecutively and in ascending order as quickly as possible. In Part B of the test, the 25 numbers are duplicated inside circles of two different colors, a sequence of pink and another of yellow. In this part, the subject must connect the consecutive numbers while alternating the color of the circles.
Behavioral effectiveness of NF on attention measures - Digit and Spatial Span | The Digit and Spatial Span tests will be assessed during the pre-treatment assessment (within three weeks before the start of the treatment) and the post-treatment assessment (within 3 weeks of the end of the treatment)
  The Spatial Span test relies on visuospatial working memory. It is a variation of the Corsi block tapping task a widely used tool in clinical neuropsychology to assess non-verbal memory deficits. The original task involves irregularly arranged mounted wooden blocks, and the examiner taps out a sequence that the patient is required to mimic. The digit span test is a very short test that evaluates a person's cognitive status that initially was part of Wechsler's Intelligence Scale. It consists of telling the participant a series of numbers and ask him to repeat them back to you in the same order you say them. The first series are composed of three numbers, the next series four numbers, then five etc. The series are repeated until one incorrect answer is observed. Both the digit and spatial span tests are frequently used in hospitals and physicians' offices in order for a clinician to quickly evaluate whether a person's cognitive abilities are normal or impaired
Behavioral effectiveness of NF on attention measures - D2-R | The D2-R test will be assessed during the pre-treatment assessment (within three weeks before the start of the treatment) and the post-treatment assessment (within 3 weeks of the end of the treatment)
  The online d2-R is the computerized version of the d2 Test of Attention - Revised. The test measures the ability to concentrate and sustain attention. It consists of picking out target symbols, from among similar symbols, under pressure of time. The participant is asked to search for and mark certain target symbols (ie., the letter "d" with two dashes). The test itself consists of 14 screens in succession, each having 60 symbols laid out in six rows of ten. All instances of "d" with two dashes are to be marked. The instruction is to work quickly, without making mistakes.
electrophysiological effectiveness of NF - EEG power and connectivity | The EEG resting state will be recorded during the pre-treatment assessment (within three weeks before the start of the treatment) and the post-treatment assessment (within 3 weeks of the end of the treatment)
  EEG analyses are based on the recording of EEG signal, which is the sum of neuronal activity, mainly post-synaptic, represented on a time axis. Based on EEG we will be able to perform analyses on qEEG, connectivity between regions. We will use BrainVision system for EEG recording of 15 minutes of resting state.
electrophysiological effectiveness of NF - P300 ERP | The P300 will be assessed during the pre-treatment assessment (within three weeks before the start of the treatment) and the post-treatment assessment (within 3 weeks of the end of the treatment)
  The P300 is a component of an event-related potential (ERP), which is a measurable brain response to a specific stimulus. It typically occurs around 300 milliseconds after the presentation of a stimulus that is unexpected, infrequent, or relevant. It is often used in cognitive neuroscience to study attention and decision-making processes. It is detected using EEG and often uses tasks like the "oddball paradigm," where subjects are asked to detect infrequent target stimuli among frequent non-targets, to elicit the P300 response.
  P300 will be assessed with an auditory oddball paradigm built using Eprime and Brain Vision EEG system.

SECONDARY OUTCOMES:
Motivation of NF training compared to standard cognitive rehabilitation | The IMI questionnaire will be provided to participants post-intervention (within 3 weeks of the end of the treatment)
  The Intrinsic Motivation Inventory (IMI) is a multidimensional measurement device intended to assess participants' subjective experience related to a target activity in laboratory experiments. It is composed of several subscales that measure enjoyment, perceived competence, effort, value, felt pressure, perceived choice. The interest/enjoyment subscale is the self-report measure of intrinsic motivation. Although research has showed that the order in which the subscales are presented is negligible, all subscales are rarely administered and researchers generally choose the subscales relevant to their study. In the present study we will administer the items related to the interest/enjoyment subscale.
Transfer to daily life and perceived effectiveness - PGIC | The PGIC questionnaire will be provided to participants post-intervention (within 3 weeks of the end of the treatment)
  The Patient's Global Impression of Change is a short questionnaire composed of two questions about the patient's perception of change related to his/her symptoms. One question is rated 1 to 7 (Likert scale) and the other one is rated 0 to 10.
Transfer to daily life and perceived effectiveness - Moss | The Moss attentional questionnaire will be provided to participants post-intervention (within 3 weeks of the end of the treatment)
  The Moss Attentional Scale was developed by Whyte and Hart to provide a reliable, quantitative and ecologically valid measure of attention-related behaviors. It is composed of 22 items, each being a descriptor rated on a five-point Likert-type scale according to how well that behavior describes the patient, ranging from "definitely true" to "definitely false."
Transfer to daily life and perceived effectiveness - GAS | The GAS questionnaire will be provided to participants post-intervention (within 3 weeks of the end of the treatment)
  The Goal Attaintment Scale (GAS) was first introduced in the 1960s by Kirusek and Sherman for assessing outcomes in mental health settings. It is a method of scoring the extent to which patients' individual goals are achieved in the course of intervention. Traditional standardised measures include a standard set of tasks (items) each rated on a standard level. In GAS, tasks are individually identified to suit the patient, and the levels are individually set around their current and expected levels of performance.

CONTACTS AND LOCATIONS:
Locations (2):
- Spain (2):
  - Irenea Neurorhb Sl, Valencia, Province de Valence
  - Servicio de Neurorrehabilitación y Daño Cerebral de los Hospitales NISA, Valencia, Spain

IPD SHARING:
Plan to Share IPD: No
Outcome and demographical/clinical data will not be made openly available as it is sensitive data and cannot be shared on open access unrestricted platforms. This is for legal reasons due to the fact that data might allow patient's identity to be revealed. Behavioural and raw EEG data (without any demographical and clinical information) might be shared with other scientists privately on platforms such as ResearchGate upon reasonable requests.

REFERENCES:
- See also: Related Info — https://irenea.es/irenea-servicio-de-neurorrehabilitacion/proyectos-internacionales/nemore/